CLINICAL TRIAL: NCT01248780
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Golimumab in the Treatment of Chinese Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: Study of Subcutaneous Golimumab in Chinese Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015913; C0524T28 (Other: Centocor)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; injection; golimumab; simponi
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Golimumab + methotrexate (MTX) (Experimental): Participants will receive golimumab 50 mg as subcutaneous (SC) (under the skin) injections administered every 4 weeks for up to 48 weeks. In addition, participants will receive a stable dose of MTX.
  Interventions: Drug: Golimumab; Drug: Methotrexate (MTX)
- Placebo + methotrexate (MTX) (Experimental): Participants will be administered Placebo SC injections at Weeks 0, 4, 8, 12, 16, and Week 20 followed by golimumab 50 mg SC injections at Week 24 and every 4 weeks thereafter through Week 48. In addition, participants will receive a stable dose of MTX.
  Interventions: Drug: Placebo; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Golimumab — 50 mg subcutaneous (SC) injection every 4 weeks for up to 48 weeks
  Arms: Golimumab + methotrexate (MTX)
Drug: Placebo — Placebo SC injections at Weeks 0, 4, 8, 12, 16, and Week 20 followed by golimumab 50 mg SC injections at Week 24 and every 4 weeks thereafter up to Week 48.
  Arms: Placebo + methotrexate (MTX)
Drug: Methotrexate (MTX) — A stable dose of MTX (oral or injectable) will be administered to participants according to the local prescribing guidelines for up to 48 weeks.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of golimumab in Chinese patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Golimumab is a type of tumor necrosis factor (TNF)-inhibitor. TNF is a naturally occurring substance in the body, and this substance may cause long-term inflammation. Golimumab may help fight disease by blocking the activity of TNF in the body and reducing inflammation and pain. Each patient who is allowed to join the study will be put into a group randomly, like flipping a coin. Patients may get either golimumab or placebo (which looks like the drug being studied but has no active ingredients, for example a sugar pill). The chance that the patient will get golimumab is 1 to 1, a 50% chance to receive golimumab and a 50% chance to receive placebo. If the patient does not have an improvement in their joints at the Week 16 visit compared to when they entered the study, and are in Group 1 (placebo group), the patient will receive golimumab 50 mg every 4 weeks starting at Week 16. If the patient is in Group 2 (golimumab 50 mg), the patient will continue to receive golimumab every 4 weeks starting at Week 16. If the patient is in Group 1 and is still receiving placebo injections, because there was improvement in their joints at Week 16, the patient will receive golimumab 50 mg every 4 weeks starting from Week 24. If the patient is in Group 2 (golimumab 50 mg) or is already receiving golimumab injections at week 24, the patient will continue to receive golimumab every 4 weeks. Safety will be monitored throughout the study, including drawing blood and looking at laboratory tests, vital signs (e.g., blood pressure), and the frequency and type of adverse events (side effects). The patient will be in the study approximately 56 weeks. Patients will receive placebo or active compound (golimumab 50 mg subcutaneous injections) every four weeks from randomization (Week 0) until Week 48.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of rheumatoid arthritis for at least 6 months

* Be on a stable dose of methotrexate for 4 weeks
* Have at least 4 swollen and 4 tender joints

Exclusion Criteria:

* Prior exposure to biologic anti-TNFalpha agents
* Inflammatory diseases other than rheumatoid arthritis
* Treatment with Disease Modifying Anti-rheumatic drug (DMARDs)/systemic immunosuppressives other than methotrexate during the 4 weeks prior to the first administration of study agent
* History of, or ongoing, chronic or recurrent infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (9):
- China (9):
  - Beijing
  - Chengdu
  - Hefei
  - Jinan
  - Nanjing
  - Shanghai
  - Suzhou
  - Wuhan
  - Xi'an

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this trial, 264 participants were randomly assigned to the 2 treatment arms.
Groups:
- Group I: Placebo + MTX -> Golimumab 50 mg + MTX: Placebo SC injections every 4 weeks from Week 0 to Week 20 (unless early escape at Week 16); golimumab 50 mg SC injections every 4 weeks from Week 16 to Week 48 if early escape; golimumab 50 mg SC injections every 4 weeks from Week 24 to Week 48 if not early escape. In addition, participants received a stable dose of methotrexate (MTX) capsules (>= 7.5 mg/week and <= 20 mg/week).
- Group II: Golimumab 50 mg + MTX: Golimumab 50 mg SC injections every 4 weeks from Week 0 to Week 48; In addition, participants received a stable dose of methotrexate (MTX) capsules (>= 7.5 mg/week and <= 20 mg/week).
Period: Overall Study
Arm/Group | Group I: Placebo + MTX -> Golimumab 50 mg + MTX | Group II: Golimumab 50 mg + MTX
Started | 132 | 132
Completed | 123 | 117
Not Completed | 9 | 15
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 2 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Not treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo + MTX -> Golimumab 50 mg + MTX | Group II: Golimumab 50 mg + MTX | Total
Number analyzed (Participants) | 132 | 132 | 264
Age Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.16) | 47.7 (11.46) | 47.2 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 110 | 214
  Male | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response, Using CRP (C-reactive Protein), at Week 14
Description: ACR 20 response is defined as >= 20% improvement in rheumatoid arthritis (RA) symptoms and disease activity.
Time Frame: Week 14
Population: Participants randomized (ie, intent-to-treat population) according to their assigned treatment group regardless of whether or not they received the assigned treatment.
Measure: Number; unit: Number of participants
Groups:
- Group I: Placebo + MTX: Placebo SC injections every 4 weeks from Week 0 to Week 20 (unless early escape at Week 16); golimumab 50 mg SC injections every 4 weeks from Week 16 to Week 20 if early escape; In addition, subjects received a stable dose of methotrexate (MTX) capsules (>= 7.5 mg/week and <= 20 mg/week).
- Group II: Golimumab 50 mg + MTX: Golimumab 50 mg SC injections every 4 weeks from Week 0 to Week 20; In addition, subjects received a stable dose of methotrexate (MTX) capsules (>= 7.5 mg/week and <= 20 mg/week).
Arm/Group | Group I: Placebo + MTX | Group II: Golimumab 50 mg + MTX
Number analyzed (Participants) | 132 | 132
Number of participants | 21 | 54
Statistical Analysis 1: Comparison: Group I: Placebo + MTX vs Group II: Golimumab 50 mg + MTX; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Disease Activity Index Score (DAS 28) Response, Using CRP (C-reactive Protein)
Description: DAS28 using CRP is a measure of tender and swollen joints (28 joints each) and the patient's assessments of disease activity. A score of higher than 5.1 indicates high disease activity, and a score below 3.2 indicates low disease activity. A DAS28 (using CRP) responder is defined as a participant with a DAS28 response of "Good" or "Moderate" at Week 14. A "Good" response is defined as a patient with a DAS28 score of <= 3.2 at Week 14 with improvement from Baseline in DAS28 score of > 1.2. A "Moderate" response was defined as a patient with DAS28 score of >3.2-5.1 at Week 14 with improvement from baseline in DAS28 score of >0.6 to >1.2 The table below shows the number of participants in each treatment group who were DAS28 responders at Week 14.
Time Frame: Week 14
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Group I: Placebo + MTX | Group II: Golimumab 50 mg + MTX
Number analyzed (Participants) | 132 | 132
Number of participants | 40 | 86
Statistical Analysis 1: Comparison: Group I: Placebo + MTX vs Group II: Golimumab 50 mg + MTX; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: American College of Rheumatology 20 Response, Using CRP, at Week 24
Description: ACR 20 response is defined as >= 20% improvement in rheumatoid arthritis (RA) symptoms and disease activity.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Group I: Placebo + MTX | Group II: Golimumab 50 mg + MTX
Number analyzed (Participants) | 132 | 132
Number of participants | 21 | 56
Statistical Analysis 1: Comparison: Group I: Placebo + MTX vs Group II: Golimumab 50 mg + MTX; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: HAQ (Disability Index of the Health Assessment Questionnaire) Score Change From Baseline
Description: The HAQ assesses the degree of difficulty a person has in accomplishing tasks in 8 categories (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). The full range of the HAQ scale is 0-24 with 0 being the best possible outcome. The HAQ score is calculated as the sum of the category scores divided by the number of categories scored, giving a possible range of scores from 0 to 3 with 0 being the best possible outcome (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, or 3=unable to do). The mean change from baseline at Week 24 in HAQ score is provided below for each treatment group. A negative change from baseline is indicative of a lesser degree of difficulty in accomplishing tasks assessed in the HAQ.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group I: Placebo + MTX | Group II: Golimumab 50 mg + MTX
Number analyzed (Participants) | 132 | 132
Scores on a scale | 0.1525 (0.69164) | -0.2623 (0.56767)
Statistical Analysis 1: Comparison: Group I: Placebo + MTX vs Group II: Golimumab 50 mg + MTX; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: 4 patients in Group I received placebo only and are not included in the safety analysis set at Week 56. 1 patient in group 2 did not receive any treatment (see participant flow) and is not included in the safety analysis set at Week 56.
Groups:
- Group I: Placebo + MTX -> Golimumab 50 mg + MTX: Placebo SC injections every 4 weeks from Week 0 to Week 12 and early escaped to receive golimumab 50 mg SC injections every 4 weeks from Week 16 to Week 48; or placebo SC injections every 4 weeks from Week 0 to Week 20 and crossed over to receive golimumab 50 mg SC injections every 4 weeks from Week 24 to Week 48. In addition, participants received a stable dose of methotrexate (MTX) capsules (>= 7.5 mg/week and <= 20 mg/week).
Arm/Group | Group I: Placebo + MTX -> Golimumab 50 mg + MTX | Group II: Golimumab 50 mg + MTX
Serious Adverse Events (participants affected / at risk) | 4/128 | 8/131
Other Adverse Events (participants affected / at risk) | 40/128 | 35/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo + MTX -> Golimumab 50 mg + MTX (N=128) | Group II: Golimumab 50 mg + MTX (N=131)
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo + MTX -> Golimumab 50 mg + MTX (N=128) | Group II: Golimumab 50 mg + MTX (N=131)
Upper Respiratory Tract Infection (Infections and infestations) | 32 | 25
Liver Function Test Abnormal (Investigations) | 7 | 8
Anaemia (Blood and lymphatic system disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days